CLINICAL TRIAL: NCT00331162
Title: Alemtuzumab Versus Thymoglobulin Induction Therapy in Kidney and Pancreas Transplantation
Brief Title: Study of Alemtuzumab Versus Anti-thymocyte Globulin to Help Prevent Rejection in Kidney and Pancreas Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BG04-498
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Graft Rejection
Keywords: Renal Transplantation; Pancreas Transplantation; Graft Rejection; Immunosuppression; Kidney failure, chronic; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Alemtuzumab; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Alemtuzumab
  Interventions: Drug: Alemtuzumab
- 2 (Active Comparator): Anti-Thymocyte Globulin
  Interventions: Drug: Anti-Thymocyte Globulin

INTERVENTIONS:
Drug: Alemtuzumab — 30 mg/100ml NS intraoperatively. Start after dexamethasone administration and prior to reperfusion of the allograft. Infuse over a minimum of 2 hours.
  Arms: 1
Drug: Anti-Thymocyte Globulin — 1.5 mg/kg per dose through a central line intraoperatively and on POD# 2 and 4, then continue on alternate days until a therapeutic tacrolimus(or cyclosporine) level is achieved, or until the SCr < 3-4 mg/dL.
  Give first dose over 6 hours, subsequent doses over 4 hours.
  Premedication to be given with the first 3 doses:
  Tylenol 650mg PO/PR Benadryl 25-50mg PO/IV Daily scheduled corticosteroid dose or other corticosteroid as deemed appropriate.
  Hold infusion if temperature > 100.5ºF; Adjust dose for low WBC or Plt count Peripheral Thymoglobulin administration: Prepare dose in 500cc NS; Add heparin 1,000 units and hydrocortisone 20mg to the bag; Infuse over a minimum of 6 hours
  Arms: 2

SUMMARY:
The purpose of this research study is to compare the effects of the two most commonly used anti-T cell induction agents(alemtuzumab and rabbit anti-thymocyte globulin) to prevent rejection in kidney and pancreas transplant patients. Alemtuzumab is Food and Drug Administration (FDA) approved for treating a certain type of cancer (leukemia), and Thymoglobulin® (rabbit anti-thymocyte globulin) is approved for anti-rejection treatment, but neither drug is FDA approved for administration at the time of transplantation to help prevent rejection. Even so, many transplant centers use these medications at the time of transplantation and believe that their use helps to decrease the risk of developing rejection following kidney and pancreas transplantation. Which drug might be better is not known. Subjects will receive either alemtuzumab (one administration) or rabbit anti-thymocyte (3 to 7 doses) at and within the first week of transplantation. Subjects will be assigned to either the alemtuzumab or rabbit anti-thymocyte globulin groups by chance. The two groups will be compared to see if there are meaningful differences for survival, organ function, side effects, and quality of life. The follow-up care after transplant for subjects in the study is the same as that for patients who are not in the study, except that a quality of life questionnaire (estimated to take 10 minutes to complete) will be completed at the time of transplant and through year 2 during selected scheduled clinic visits. A retrospective chart review will occur at 3-5 years post-transplant to follow incidence of chronic rejection, patient and graft survival and graft function.

DETAILED DESCRIPTION:
Anti-Thymocyte Globulin, rabbit (r-ATG, Thymoglobulin®) is a polyclonal antibody against T-lymphocytes that is used for the prevention and treatment of acute allograft rejection. r-ATG induction therapy is effective in preventing acute allograft rejection, however the usual 7-14 day course involves extensive clinical monitoring and is costly. Recent studies had suggested that smaller cumulative doses are efficacious for induction therapy, and may have an advantage by decreasing the adverse effects associated with the agent (such as leukopenia and thrombocytopenia). Our program subsequently modified our r-ATG induction regimen in November 2001 to give doses on alternate days for at least three doses and has achieved excellent results. However, this regimen is somewhat complex in that it requires central venous access for administration, pre-medication administration to prevent infusion-related reactions, and monitoring of vital signs during each infusion.

Alemtuzumab (Campath®) is a humanized monoclonal antibody to CD52 that is FDA approved for the treatment of B-cell chronic lymphocytic leukemia (B-CLL), but has also been used for immunosuppression induction at the time of solid organ transplant and as anti-rejection therapy. CD52 is present on most lymphocytes, macrophages, monocytes, and NK cells, and causes antibody-dependent cell lysis following the binding of alemtuzumab to the CD52 surface antigen. Alemtuzumab produces significant lymphocyte depletion similar to r-ATG, so some investigators began evaluating it as a preconditioning agent in tolerance protocols (using very low-dose maintenance immunosuppression) in solid organ transplantation. While these studies showed no significant tolerogenic potential for alemtuzumab, one or two 20-30 mg doses of alemtuzumab produced a similar degree of lymphocyte depletion as r-ATG administration. Based on these preliminary data in transplant recipients and prior safety data obtained from safety and efficacy studies of alemtuzumab in patients with rheumatoid arthritis, some US transplant centers changed from using r-ATG to alemtuzumab as their primary induction agent. Most of these centers (notably Wisconsin and Northwestern, where more than 500 kidney and pancreas patients have received alemtuzumab, personal communication Dixon Kaufman, Northwestern) use one or two doses of alemtuzumab for induction, followed by a traditional 2-3 drug maintenance immunosuppressive regimen (rather than the low-dose immunosuppression used in the tolerance protocols).

Knechtle and colleagues from the University of Wisconsin have reported a comparable incidence of acute rejection and favorable graft survival in 130 patients who received a single intraoperative 30 mg dose (+/- an additional dose on post-operative day 1) of alemtuzumab compared with a historical cohort who received r-ATG, OKT3, an IL-2 receptor antagonist, or no induction. In addition, the group found that there was a dramatically lower incidence of acute rejection in the patients who experienced delayed graft function in the alemtuzumab group (9% vs 45% in the control group, p=0.0078).

The use of alemtuzumab as an induction agent in solid organ transplantation is appealing. Only a single intraoperative dose would be required (compared with between 2 and 6 additional doses of r-ATG post-op), thereby eliminating the necessity for central venous access and extensive clinical and nurse monitoring. In addition, the cost of therapy would be less with alemtuzumab than with r-ATG. At WFUBMC, 18 recipients of kidney or kidney/pancreas transplants who received alemtuzumab have had only a 9% six-month rejection rate. Our clinical experience suggests that the agents produce similar results; however, a prospective, randomized study to compare the safety and efficacy of alemtuzumab with r-ATG has not been reported. Also, although alemtuzumab would offer a significant medication cost savings over r-ATG, the impact on the overall cost of care has yet to be established. A comparative study will help us decide if we should make alemtuzumab our new standard of care at this institution.

The purpose of this study is to evaluate the use of alemtuzumab (Campath-1H) for induction therapy in kidney and pancreas transplantation compared to our standard of care, alternate-day r-ATG.

ELIGIBILITY:
Enrollment of kidney transplant patients has been completed. The protocol has been amended to enroll 50 additional subjects who will receive either a simultaneous pancreas and kidney transplant, pancreas after kidney transplant, or solitary pancreas transplant.

Inclusion Criteria:

* Male or female patients who receive a simultaneous pancreas and kidney transplant, pancreas after kidney transplant, or solitary pancreas transplant
* Age 18 to 65
* Females of child bearing potential must have a negative pregnancy test at time of transplant
* Ability to give informed consent

Exclusion Criteria:

* Inability to give informed consent
* ABO incompatibility
* T-cell or B-cell positive cross match
* Patients with a previous hypersensitivity to alemtuzumab, anti-thymocyte globulin, or any monoclonal or polyclonal antibody preparation
* Current active infection (currently receiving antibiotics, treatment for active infection within 1 week of transplant, or medical judgement)
* Hepatitis B surface antigen positive
* Human immunodeficiency virus positive
* Any malignancy within 2 years except for successfully treated basal or squamous cell carcinoma of skin
* Pregnancy
* Breast feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2005-02 (Actual); Primary Completion 2011-11-28 (Actual); Study Completion 2011-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Farney, MD, Ph.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brennan DC, Flavin K, Lowell JA, Howard TK, Shenoy S, Burgess S, Dolan S, Kano JM, Mahon M, Schnitzler MA, Woodward R, Irish W, Singer GG. A randomized, double-blinded comparison of Thymoglobulin versus Atgam for induction immunosuppressive therapy in adult renal transplant recipients. Transplantation. 1999 Apr 15;67(7):1011-8. doi: 10.1097/00007890-199904150-00013. PMID 10221486
- [Background] Knechtle SJ, Pirsch JD, H Fechner J Jr, Becker BN, Friedl A, Colvin RB, Lebeck LK, Chin LT, Becker YT, Odorico JS, D'Alessandro AM, Kalayoglu M, Hamawy MM, Hu H, Bloom DD, Sollinger HW. Campath-1H induction plus rapamycin monotherapy for renal transplantation: results of a pilot study. Am J Transplant. 2003 Jun;3(6):722-30. doi: 10.1034/j.1600-6143.2003.00120.x. PMID 12780564
- [Background] Kaufman DB, Leventhal JR, Gallon LG, Parker MA. Alemtuzumab induction and prednisone-free maintenance immunotherapy in simultaneous pancreas-kidney transplantation comparison with rabbit antithymocyte globulin induction - long-term results. Am J Transplant. 2006 Feb;6(2):331-9. doi: 10.1111/j.1600-6143.2005.01166.x. PMID 16426317
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Started | 113 | 109
Completed | 113 | 109
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin | Total
Number analyzed (Participants) | 113 | 109 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12) | 49 (13) | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 47 | 93
  Male | 67 | 62 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 36 | 70
  White | 74 | 69 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Patient Survival
Description: The number of patients that survived after transplantation occurred was reported.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 113 | 109
Participants | 109 | 104

2. Primary Outcome: Graft Survival
Description: The number of patients with graft survival after kidney alone, simultaneous pancreas-kidney (SPK), and pancreas after kidney (PAK) transplant.
Time Frame: 5 years
Population: Number the analyzed in one or more rows differs from overall number analyzed because there were subgroups for transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 113 | 109
Participants
  Kidney alone: number analyzed (Participants) | 85 | 95
  Kidney alone | 78 | 84
  SPK: number analyzed (Participants) | 24 | 14
  SPK | 21 | 13
  PAK: number analyzed (Participants) | 4 | 0
  PAK | 4 | 0

3. Primary Outcome: Acute Rejection
Description: The number of patients with acute rejection after transplantation was reported.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 113 | 109
Participants | 16 | 28

4. Secondary Outcome: Hematologic Adverse Events
Time Frame: 2 years
Population: No data was collected
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Infectious Adverse Events
Description: Number of events for infectious adverse events were reported (Polyoma virus nephropathy (PVD), cytomegalovirus (CMV), bacterial and fungal infections).
Time Frame: 2 years
Measure: Number; unit: number of events
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 113 | 109
number of events
  CMV | 9 | 18
  PVN | 1 | 8
  Fungal infections | 11 | 11
  Bacterial Infections | 89 | 92

6. Secondary Outcome: Other Adverse Events
Description: Number of patients with other adverse events (posttransplant lymphoproliferative disorder (PTLD), and nonskin malignancy), were reported.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 113 | 109
Participants
  PTLD | 0 | 1
  Other Nonskin Malignancy | 0 | 2

7. Secondary Outcome: Cost
Time Frame: 2 years
Population: No data was collected
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Health Status and Quality of Life
Time Frame: 2 years
Population: No data was collected.
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Alemtuzumab | Anti-Thymocyte Globulin
All-Cause Mortality (participants affected / at risk) | 4/113 | 5/109
Serious Adverse Events (participants affected / at risk) | 11/113 | 44/109
Other Adverse Events (participants affected / at risk) | 0/113 | 0/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab (N=113) | Anti-Thymocyte Globulin (N=109)
Cardiovascular Disease (Cardiac disorders) | 2 | 2
Renal Allograft Pseudoaneurysm (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Blood and lymphatic system disorders) | 0 | 1
Posttransplant lymphoproliferative disorder (Blood and lymphatic system disorders) | 0 | 1
Fungal Infection (Infections and infestations) | 11 | 11
Viral Infections (Infections and infestations) | 10 | 27
Other (nonskin) Malignancy (Blood and lymphatic system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes